CLINICAL TRIAL: NCT07151963
Title: Effects of Prolonged Continuous Theta Burst Stimulation in Chemotherapy-induced Peripheral Neuropathy: a Randomized Cross- Over Trial
Brief Title: Effects of Prolonged Continuous Theta Burst Stimulation in Chemotherapy-induced Peripheral Neuropathy
Acronym: CIPN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13-IRB009
Record Dates: First submitted 2025-08-18; First posted 2025-09-03 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Females
Keywords: conventional repetitive transcranial magnetic stimulation; breast cancer; chemotherapy induced peripheral neuropathy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prolonged continuous TBS (pcTBS) (Experimental): pcTBS over M1
  Interventions: Device: prolonged continuous TBS
- 20 Hz rTMS (Active Comparator): 20 Hz rTMS over M1
  Interventions: Device: 20 Hz rTMS

INTERVENTIONS:
Device: prolonged continuous TBS — prolonged continuous theta burst stimulation
  Arms: prolonged continuous TBS (pcTBS)
Device: 20 Hz rTMS — 20 Hz repetitive transcranial magnetic stimulation
  Arms: 20 Hz rTMS

SUMMARY:
Laboratory studies have shown that prolonged continuous theta burst stimulation (pcTBS) provides better pain relief than 10 Hz repetitive transcranial magnetic stimulation (rTMS), with a shorter stimulation time, making it more practical for clinical use. Chemotherapy-induced peripheral neuropathy often causes neuropathic pain in cancer patients. The aims of this study are:

1. To compare the effects of pcTBS and 20 Hz rTMS on chemotherapy-induced peripheral neuropathy;
2. To compare the effects of pcTBS applied to the primary motor cortex versus the dorsolateral prefrontal cortex on neuropathic pain as well as depression and anxiety.

DETAILED DESCRIPTION:
**Phase 1:** Investigators will recruit 20 breast cancer patients who have chemotherapy-induced peripheral neuropathy. They will be randomly divided into two groups.

* Group 1 will first receive pcTBS. After an 8-week break, they will then receive 20 Hz rTMS.
* Group 2 will receive the treatments in the opposite order.

Each treatment lasts for 5 consecutive days. Before and after each treatment, patients will be assessed using:

* A pain visual analog scale (to measure pain levels)
* A Neuropathic Pain Symptom Inventory (The scale ranges from zero to 10, with zero indicating no pain at all and 10 indicating the worst imaginable pain)

  • * A Depression Anxiety Stress Scale 21 (The scale ranges from 0-63, with a higher scores mean a worse outcome)

  o * Clinical pressure pain threshold tests (Higher PPT values indicate a higher tolerance to pressure pain (less sensitivity).
* Nerve conduction studies **Phase 2:** Another 20 breast cancer patients with chemotherapy-induced peripheral neuropathy will be recruited and randomly divided into two groups.
* Group 1 will first receive pcTBS on the primary motor cortex. After an 8-week break, they will receive the same stimulation on the left dorsolateral prefrontal cortex.
* Group 2 will receive the treatments in the opposite order.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients aged between 18- and 80-years-old with CIPN
* history of receiving chemotherapy including taxane-based neurotoxic agents
* with neuropathic pain, score≥3 in a 0-10 VAS pain scale.
* with fair cognition and can cooperate to evaluate pain severity.
* neither at end-stage cancer nor at the estimated survival time less than 6 months.

Exclusion Criteria:

* brain tumor or history of epilepsy
* intracranial metallic devices, artificial cochleae, pacemakers, or any other metal device
* recent myocardial ischemia or unstable angina
* severe cognitive dysfunction or pregnancy
* injuries or fractures in the part of neuropathic pain

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
visual analogue pain scale (VAS pain scale) | baseline, pre-intervention and immediately after completion the intervention and at 4 weeks follow-up
  visual analogue pain scale (VAS) range from 0-100, with a higher score inducating more pain

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale 21 | baseline and after completion the intervention and at 4 weeks follow-up
  Depression Anxiety Stress Scale 21 scale ranges from 0-63, with a higher scores mean a worse outcome.
pressure pain threshold test | baseline and after completion the intervention and at 4 weeks follow-up
  o Higher pressure pain threshold values indicate a higher tolerance to pressure pain (less sensitivity).
Neuropathic Pain Symptom Inventory | baseline and after completion the intervention and at 4 weeks follow-up
  Neuropathic Pain Symptom Inventory ranges from zero to 10, with zero indicating no pain at all and 10 indicating the worst imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Shiung Horng, MD., PhD., Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
confidential data